CLINICAL TRIAL: NCT05853302
Title: Outcome and Cost-effectiveness of Robot-assisted vs Laparoscopic Lateral Transabdominal Adrenalectomy
Brief Title: Robot-assisted vs Laparoscopic Lateral Transabdominal Adrenalectomy
Acronym: RvsL-TLA
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4853
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2023-02

CONDITIONS: Adrenalectomy; Status
Keywords: minimally-invasive surgery; robotic surgery; lateral transabdominal adrenalectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Laparoscopic TLA: Patients who underwent laparoscopic lateral transabdominal unilateral adrenalectomy
- Robotic TLA: Patients who underwent robotic lateral transabdominal unilateral adrenalectomy

SUMMARY:
This retrospective study evaluates the safety and the effectiveness of robotic adrenalectomy when compared to laparoscopic approach in patients who underwent minimally-invasive lateral transperitoneal unilateral adrenalectomy

DETAILED DESCRIPTION:
During the last twenty years, minimally-invasive surgery became the first choice for the surgical treatment of most of adrenal diseases. The advantages of minimally-invasive techniques are mostly to relate to the significative post-operative morbidity reduction. Adrenalectomy is a technical demanding procedure, requiring a cautious and precise dissection in the retroperitoneal space, so that endoscopic magnification may represent an essential tool. Several minimally-invasive approaches to adrenalectomy have been described, including anterior and lateral laparoscopic or lateral and posterior retroperitoneal techniques. Lateral transabdominal approach is the most frequently used for robotic adrenalectomy. However, routinary use of robotic platforms is limitated by their high costs.

Laparoscopic adrenalectomy was described by Gagner at al. in 1992, by means of a lateral transperitoneal approach. Several retrospective studies showed the advantages of laparoscopic approach compared to laparotomic procedure, such as lower post-operative pain, morbidity and hospital stay. Lateral transabdominal laparoscopic adrenalectomy is nowadays the most frequently used technique. One of the main advantages is related to the possibility of using the gravity effect during surgical dissection. Indeed, after the mobilization of the anatomic structures next to the adrenal gland (liver on the right side and splenopancreatic block on the left side), no more manipulations are necessary during the procedure. Moreover, this approach guarantees a wide working space, with the exposure of conventional anatomic landmarks, allowing an adequate vascular control. A further advantage consists in the possibility of exploring the whole abdominal cavity, therefore permitting the treatment of other surgical clinical conditions. Technically speaking, the main condition for the procedure success is a complete knowledge of surgical anatomy and an adequate surgical expertise, so that different approaches may be chosen basing on both patients' and lesions' features.

In 1999 Piazza et al. and Hubens et al. described robotic approach to adrenalectomy by means of AESOP 2000 platform. Then, "Da Vinci" platform (Intuitive Surgical, Sunnyvale, CA, USA) was introduced in clinical practice. After that, robotic adrenalectomies have been performed in several centers, proving the safety and feasibility of such procedure. "Da Vinci" platform allowed to maintain the same advantages of minimally-invasive approaches, with a reduction of the difficulties due to their technical limitations. Indeed, ergonomic superiority, tridimensional vision, tremors reduction and major freedom degrees related to the robotic instruments allow an easier surgical dissection.

Minimally-invasive adrenalectomy is the gold standard for the treatment of <6 cm adrenal lesions. Feasibility of endoscopic adrenalectomy for the treatment of wider or suspected for malignancy adrenal lesions still remains debated. National Institute of Health (NIH) Position Statement showed that adrenal cortical carcinoma prevalence is directly related to the lesion diameter, representing 2% of <4 cm lesions, 6% of 4,1-6 cm lesions and 25% of >6 cm lesions. However, lesion diameter alone is a too aspecific factor to be considered the parameter of choice of the surgical approach. Indeed, about 75% of >6 cm adrenal lesions result benign after definitive histological examination. Furthermore, several works in literature showed that the oncologic radicality of minimally-invasive approaches to localized malignant lesions is not inferior comparing to conventional laparotomic procedures. However, European Society of Endocrine Surgeon (ESES) and European Network for the Study of Adrenal Tumors (ENSAT) for the treatment of adrenal lesions suggest that transperitoneal approach should be the procedure of choice to guarantee optimal intraoperative stadiation, complete oncologic resection, capsular effraction risk and verify loco-regional structures infiltration.

Most studies demonstrated that TLA is a safe and effective procedure with low morbidity and mortality rates. Post-operative complications rates are not easy to interpretate due to the lack of standardization among the studies, though their range could be assessed between 2.9 and 15.5%. Complications and conversions risk factors, such as surgeon's expertise and center's volume, patient's anatomical characteristics and lesion's features, have been evaluated in monocentric and multicentric studies. More precisely, volume center and surgical expertise impact on clinical outcome have been demonstrated in several studies. Park et al. published a retrospective analysis of 344 adrenalectomies and documented a major complications rate (18.3 vs 11.3%) and a longer hospital stay (5.5 vs 3.9 days) in those procedures performed in center with low volume. Also, Palazzo et al. showed a significative increase in hospital stay and readmission within 30 days in low volume centers. Bergamini et al. identified age, BMI, lesion diameter and catecholaminergic secretion as risk factors for complications, with low complications rates in referral centers.

Among patients' characteristics, the major risk factors for complications and conversions were obesity, history of abdominal surgery, lesion side, patients comorbidity and catecholaminergic secretion. Obesity (BMI≥30 Kg/m2) has been reported as a risk factor for post-operative complications. However, more recently such conditions turned to be associated only to an operative time increasing. History of abdominal surgery has been also reported as a risk factor for intra- and post-operative complications. However, recent case series proved that TLA performed after previous abdominal surgery did not lead to major conversion and complications rates. Lesion diameter has been evaluated in several experiences as complications risk factor, with different dimensional cut-off. An higher post-operative complications rate have been reported in patients with lesions >60 mm. However, other studies with different cut-off (60-80 mm) did not confirm such results.

To date, conversion rate to laparotomic surgery set to a median of 2%, with a range of 0-13%. Vascular and organs' lesions, as well as the technical difficulties, are the most frequent causes of conversion.

The TLA-related reported mortality is 0-0.8%. The most frequent causes of death are massive bleeding, pancreatitis, pulmonary embolism and sepsis.

Systematic reviews and meta-analysis showed the safety and effectiveness of the robotic approach to adrenalectomy. The reported operative times are different among the published works in literature, with median values of 98-234 minutes. Brunaud et al. identified some criteria that might influence the operative times, such as surgeon's expertise, the assistant training level, lesion diameter (with lower times in case of lesion<45 mm). Longer operative times are tipically associated with the beginning of the surgical experience and may be related to the docking. However, in referral centers with high experience in endoscopic adrenal surgery, docking times are significantly reduced after the learning curve is completed. In our experience, docking time requires about 10 minutes to be completed. Blood loss and hospital stay length are generally considered comparable to TLA. However, several authors report less blood loss and shorter hospital stay in case of robotic adrenalectomy. Robotic surgery conversion rates to the laparoscopic and laparotomic approach vary between 0% - 40% and 0% - 10%, respectively. Conversion-related conditions are adhesions, bleeding and technical difficulties. Retrospective series and meta-analysis confirmed that laparoscopic and robotic morbidity and mortality rates are comparable. High costs still represent a limitation of robotic procedures. Brunaud et al. evidenced 2.3 times higher costs for robotic approach. Total costs are proportional to total procedures per year and to instruments costs, while operative time has a marginal role. Similar results have been published by Morino et al. Some authors achieved different results, as costs analysis was influenced by the specific health system reimbursement. In De Crea et al. cost-analysis 131 patients who underwent adrenalectomy between January 2017 and September 2019 (39 PRA, 80 TLA and 12 RA) have been compared. Cost-analysis considered Italian Health system reimbursement basing on Diagnosis Related Group (DRG). All the procedures, including RA, presented positive marginality, with comparable values between PRA and TLA, superior to RA in both cases. Thoughout a subgroups analysius, marginality difference between RA and the other approaches was reduced of 20% in case of lesion >4 cm. The results confirmed that RA may present advantages in case of challenging cases, such as obese patients or large lesions.

ELIGIBILITY:
Inclusion Criteria:

Patients who underwent minimally-invasive unilateral adrenalectomy with lateral transabdominal approach between June 1st 1997 and December 31st 2021

Exclusion Criteria:

Patients who underwent bilateral or retroperitoneoscopic adrenalectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In consideration of the 15%-minimally invasive procedure-related morbidity rate (both with laparoscopic and robotic approach), the 5%-significativity, the 80%-study power and the 10%-non-inferiority limit, the sample size is 316 patients. Such sample size is divided in 15 patients per group (Sealed Envelope Ltd. 2012. Power calculator for binary outcome noninferiority trial. [Online] Available from: https://www.sealedenvelope.com/power/binary-noninferior/ [Accessed Mon Jan 31 2022]).
Sampling Method: Non-Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Post-operative complications | June 1997-December 2021
  Evaluation of post-operative complications within 30 days from adrenalectomy

SECONDARY OUTCOMES:
Mortality | June 1997-December 2021
  Evaluation of mortality rate within 30 days from adrenalectomy
Robotic procedure effectiveness | June 1997-December 2021
  Evaluation of effectiveness in terms of operative time, post-operative hospital stay and cost-analysis

CONTACTS AND LOCATIONS:
Overall Officials: Marco Raffaelli, Prof, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided